CLINICAL TRIAL: NCT05595330
Title: Effect of Lymphedema Prevention Program Based on Theory of Knowledge-attitude-practice on Postoperative Breast Cancer Patients: a Randomized Clinical Trial
Brief Title: Effect of Lymphedema Prevention Program Based on Theory of Knowledge-attitude-practice on Postoperative Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Shi Bohui, Nurse in charge, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 19900601
Record Dates: First submitted 2022-09-23; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Patients in the intervention group were managed with an upper extremity lymphedema prevention program.
  Interventions: Behavioral: Lymphedema prevention protocols
- control group (No Intervention): The control group received normal perioperative and chemotherapy nursing measures

INTERVENTIONS:
Behavioral: Lymphedema prevention protocols — Coming for surgery: A PPT lecture; 2. A seminar; 3. Patients were given a lymphedema prevention brochure; 4. Diary cards for exercise is given and instruct patients to fill out daily; 5. Establish a WeChat group.
  The first chemotherapy:1. Review diary card and provide guidance and education. 2. A PPT lecture; 3. A seminar; 4. Play functional exercise videos in the recovery room; 5. Rehabilitation volunteers come to the ward to form mutual help groups with patients under the guidance of subject team members; 6. Instruct regular exercise and avoid behaviors that can lead to lymphedema. 7. Ask about the exercise and whether there is any swelling and discomfort and give guidance.
  The second chemotherapy: 1. A PPT lecture; 2. A seminar; 3. Play functional exercise videos in the recovery room.
  The third chemotherapy: 1. Routine nursing; 2. Assess patients' knowledge of lymphedema prevention and exercise compliances; 3. Play functional exercise videos in the recovery room.
  Arms: intervention group

SUMMARY:
According to the inclusion and exclusion criteria, a total of 108 patients were enrolled and randomly divided into control group (n = 56) and intervention group (n = 52). The control group received routine nursing, while the intervention group received upper limb lymphedema prevention program for breast cancer patients after surgery. Before surgery, at the third chemotherapy (about 2.1 months after surgery) and the sixth chemotherapy (about 4.2 months after surgery), the self-designed general information questionnaire was used to investigate the patient's basic situation, and the corresponding tools were used to measure the volume of the patient's upper arm, the grip strength of the affected arm, and the range of motion of the affected shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

* Female patients were≥18 years old
* Pathological puncture confirmed breast cancer with unilateral, no recurrence, and no metastasis
* Patients with clinical TNM stageⅠ~Ⅲ
* Patients with proposed surgery and 6 or more chemotherapy
* The patient was conscious and aware of his condition, with no cognitive impairment or communication problems

Exclusion Criteria:

* Patients who had cancer other than breast cancer
* Patients who had history of arm or neck trauma, infection or surgery
* Patients who had serious diseases such as cardiovascular, cerebrovascular, liver, kidney, etc
* Patients who had upper limb disability or the affected limb has edema before surgery
* Patients who had thrombus in the blood vessels of the affected limb

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Changes in breast cancer-related lymphedema at baseline,9 weeks after surgery,and 18 weeks after surgery | Baseline-9 weeks after surgery-18 weeks after surgery
  Use an inelastic, flexible soft ruler to measure the circumference at 5 positions on the flat wrist crease, 0cm, 10cm, 20cm, 30cm, and 40cm on the wrist crease. The upper limb can be divided into 4 truncated cones, and the measured value is accurate to 0.1 cm. The upper arm volume is calculated using the formula , each h is 10 cm, C1 and C2 are the circumferences next to the two measurement points, and then add up the limb volumes at several positions to get the upper arm volume.
  According to the International Society of Lymphoma, a volume difference of 10% or more is defined as lymphedema, less than 20% is mild lymphedema, 20% - 40% is moderate lymphedema, and greater than 40% is defined as severe lymphedema.
  Change(Baseline-9 weeks after surgery-18 weeks after surgery)

SECONDARY OUTCOMES:
Changes in grip strength at baseline,9 weeks after surgery,and 18 weeks after surgery | Baseline-9 weeks after surgery-18 weeks after surgery
  The grip strength of the affected side was measured with the help of electronic grip strength meter. Test method: The patient stands straight with the arm down and the affected hand grasps the grip strength meter with force. Two measurements were taken and the average was taken.
  Change(Baseline-9 weeks after surgery-18 weeks after surgery)
Changes in Shoulder range of motion at baseline,9 weeks after surgery,and 18 weeks after surgery | Baseline-9 weeks after surgery-18 weeks after surgery
  The range of motion (ROM) of the upper limb of breast cancer patients was measured with a circular goniometer (0°-360°) . The rehabilitation technician measured the upper limb mobility in six directions: forward flexion, back extension, abduction, adduction, internal rotation, and external rotation.
  Change(Baseline-9 weeks after surgery-18 weeks after surgery)
Change in Arm disability at baseline,9 weeks after surgery,and 18 weeks after surgery | Baseline-9 weeks after surgery-18 weeks after surgery
  The Chinese version of the DASH scale, adapted from the DASH scale developed by Beaton, was used to assess the upper limb condition of the patients. Cronbach's A coefficient was 0. 911, and the intra-group correlation coefficient was 0. 882, which had good reliability and validity. The highest score is 100 and the lowest is 0, with higher scores indicating more severe upper arm problems.
  Change(Baseline-9 weeks after surgery-18 weeks after surgery)
Change in Quality of life at baseline,9 weeks after surgery,and 18 weeks after surgery | Baseline-9 weeks after surgery-18 weeks after surgery
  Quality of life was evaluated using Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer, which was developed by Cella. It was translated into Chinese by Wan and the Cronbach 'α for each sub-scale was 0.61-0.84.The questionnaire had 36 items classified into five dimensions and all the items were measured with a 5-point Likert scale, The highest score is 144 and the lowest is 0,with higher scores indicating higher levels of quality of life.
  Change(Baseline-9 weeks after surgery-18 weeks after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Xi 'an, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05595330/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT05595330/SAP_001.pdf
  • Informed Consent Form (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05595330/ICF_002.pdf